CLINICAL TRIAL: NCT00261833
Title: A Randomized, Placebo-Controlled, Double-Blind, Multicenter Phase III/IV Study to Compare the Efficacy and Safety of 60mg/kg Body Weight of Zemaira® Weekly I.V. Administration With Placebo Weekly I.V. Administration in Chronic Augmentation and Maintenance Therapy in Subjects With Emphysema Due to Alpha1-Proteinase Inhibitor Deficiency
Brief Title: Zemaira in Subjects With Emphysema Due to Alpha1-Proteinase Inhibitor Deficiency
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CE1226_4001; 1449 (Other: CSL Behring); 2005-003459-12 (EudraCT Number)
Record Dates: First submitted 2005-12-02; First posted 2005-12-05 (Estimated); Results first posted 2015-01-19 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Alpha1-proteinase Inhibitor Deficiency; Emphysema
Keywords: Alpha1-proteinase inhibitor deficiency; Emphysema; Chronic augmentation and maintenance therapy
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Emphysema | interventions — alpha 1-Antitrypsin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zemaira® (Experimental)
  Interventions: Biological: Alpha1-proteinase inhibitor
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Alpha1-proteinase inhibitor — 60 mg/kg body weight/week intravenous
  Other Names: Zemaira®
  Arms: Zemaira®
Other: Placebo — Lyophilized preparation: 60 mg/kg body weight/week intravenous
  Arms: Placebo

SUMMARY:
This is a randomized, placebo-controlled, double-blind, multicenter phase III/IV study to compare the efficacy and safety of Zemaira® with placebo in subjects with emphysema due to alpha1-proteinase inhibitor deficiency. The effect of Zemaira® on the progression of emphysema will be assessed by the decline of lung density, measured by computed tomography (CT).

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age and willing to sign informed consent.
* Males and non-pregnant, non-lactating females whose screening pregnancy test is negative and who are using contraceptives methods deemed reliable by the investigator.
* Diagnosis of alpha1-proteinase inhibitor (A1-PI) deficiency (serum A1-PI levels < 11 μM or < 80 mg/dL). This includes newly diagnosed subjects, previously untreated subjects, currently treated subjects, and subjects currently not on treatment therapy but on treatment in the past.
* Subjects with emphysema and forced expiratory volume in 1 second (FEV1) ≥ 35% and ≤ 70% (predicted).
* No signs of chronic or acute Hepatitis A, Hepatitis B, Hepatitis C or HIV infection (negative serologies for HIV and viral hepatitis). In case of positive serologies for viral hepatitis, vaccination status or negative IgM should be available.

Exclusion Criteria:

* Any relevant chronic diseases or history of relevant diseases (e.g., severe renal insufficiency) except respiratory or liver disease secondary to alpha1-proteinase inhibitor deficiency. Subjects with well-controlled, chronic diseases may be included after consultation with the treating physician and the sponsor.
* Current evidence of alcohol abuse or history of abuse of illegal and/or legally prescribed drugs such as barbiturates, benzodiazepines, amphetamines, cocaine, opioids, and cannabinoids.
* History of allergy, anaphylactic reaction, or severe systemic response to human plasma derived products, or known mannitol hypersensitivity, or history of prior adverse reaction to mannitol.
* History of transfusion reactions.
* Selective IgA deficiency.
* Acute illness within one week prior to the first administration of the investigational medicinal product (IMP). Start of treatment after recovery is possible.
* Current tobacco smoker (smoking has to be ceased at least 6 months prior study inclusion). Subjects with a positive cotinine test due to nicotine replacement therapy (e.g. patches, chewing gum) or snuff are eligible.
* Conditions or behaviors that interfere with attending scheduled study visits in the opinion of the investigator.
* History of non-compliance.
* Administration of any other experimental new drug or participation in an investigation of a marketed product within one month prior to the screening visit date.
* Inability to perform necessary study procedures.
* Lung transplantation, lung volume reduction surgery or lobectomy or being on a waiting list for any such surgeries.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2006-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Director Immonology & Pulmonology, Clinical R&D, Study Director — CSL Behring
Locations (28):
- United States (4):
  - Study Site, Denver, Colorado
  - Study Site, Miami, Florida
  - Study Site, Hershey, Pennsylvania
  - Study Site, Tyler, Texas
- Australia (6):
  - Study Site, Darlinghurst, New South Wales
  - Study Site, New Lambton, New South Wales
  - Study Site, Brisbane, Queensland
  - Study Site, Adelaide, South Australia
  - Study Site, Nedlands, Western Australia
  - Study Site, Fitzroy
- Canada (3):
  - Study Site, Vancouver, British Columbia
  - Study Site, Halifax, Nova Scotia
  - Study Site, Toronto, Ontario
- Study Site, Prague, Czechia
- Denmark (2):
  - Study Site, Aarhus
  - Study Site, Hellerup
- Study Site, Tartu, Estonia
- Study Site, Oulu, Finland
- Germany (4):
  - Study Site, Berlin
  - Study Site, Essen
  - Study Site, Heidelberg
  - Study Site, Nuremberg
- Study Site, Dublin, Ireland
- Poland (2):
  - Study Site, Krakow
  - Study Site, Warsaw
- Study Site, Bucharest, Romania
- Study Site, Barnaul, Russia
- Study Site, Malmo, Sweden

REFERENCES:
- [Derived] Greulich T, Chlumsky J, Wencker M, Vit O, Fries M, Chung T, Shebl A, Vogelmeier C, Chapman KR, McElvaney NG; RAPID Trial Group. Safety of biweekly alpha1-antitrypsin treatment in the RAPID programme. Eur Respir J. 2018 Nov 29;52(5):1800897. doi: 10.1183/13993003.00897-2018. Print 2018 Nov. PMID 30237305
- [Derived] Chapman KR, Burdon JG, Piitulainen E, Sandhaus RA, Seersholm N, Stocks JM, Stoel BC, Huang L, Yao Z, Edelman JM, McElvaney NG; RAPID Trial Study Group. Intravenous augmentation treatment and lung density in severe alpha1 antitrypsin deficiency (RAPID): a randomised, double-blind, placebo-controlled trial. Lancet. 2015 Jul 25;386(9991):360-8. doi: 10.1016/S0140-6736(15)60860-1. Epub 2015 May 27. PMID 26026936

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter, multinational study enrolled participants at 28 study centers in Europe, North America, and Australia.
Pre-assignment Details: Screening took place 1 to 4 weeks prior to the first dose of randomized investigational product (ie, either Zemaira® or placebo). A total of 208 participants were screened; 28 of these did not fulfill all eligibility criteria and were therefore screening failures.
Period: Overall Study
Arm/Group | Zemaira® | Placebo
Started | 93 | 87
Completed | 84 | 69
Not Completed | 9 | 18
Not completed — Death | 1 | 3
Not completed — Adverse Event | 1 | 4
Not completed — Withdrawal by Subject | 5 | 7
Not completed — Protocol Violation | 0 | 1
Not completed — Suspicion of pulmonary cancer | 0 | 1
Not completed — Lung transplantation | 1 | 1
Not completed — Missing reason | 1 | 0
Not completed — Not interested in being participant | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zemaira® | Placebo | Total
Number analyzed (Participants) | 93 | 87 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.81 (6.193) | 52.40 (7.812) | 53.13 (7.374)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 37 | 82
  Male | 48 | 50 | 98
Baseline percent predicted forced expiratory volume in 1 second (FEV1) [Mean (Standard Deviation); unit: percentage] | 47.4 (12.1) | 47.2 (11.1) | 47.3 (11.6)
Baseline diffusion capacity of carbon monoxide (DLCO) [Mean (Standard Deviation); unit: mL/min/mmHg] | 13.6 (5.3) | 15.0 (5.6) | 14.3 (5.5)
Number of participants with ZZ genotype (A1-PI deficiency), or SZ, Z / Null or Other genotype [Number; unit: participants]
  ZZ | 83 | 83 | 166
  SZ | 2 | 0 | 2
  Z / Null | 2 | 1 | 3
  Other | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Annual Rate of Change in Lung Density
Description: As measured by centralized, standardized computer tomographic (CT) lung densitometry. CT scans were acquired at 2 inspiration states: TLC (ie, full inspiration) and FRC (ie, full expiration). Results were adjusted for total lung volume and are presented as point estimates for the average rate of decline in each treatment group.
Time Frame: Over a 2-year period
Population: All randomized participants with at least 1 valid CT scan.
Measure: Least Squares Mean (Standard Error); unit: g/L per year
Arm/Group | Zemaira® | Placebo
Number analyzed (Participants) | 92 | 85
g/L per year
  TLC + FRC combined | -1.50 (0.22) | -2.12 (0.24)
  TLC | -1.45 (0.23) | -2.19 (0.25)
  FRC | -1.55 (0.24) | -2.02 (0.26)
Statistical Analysis 1: Comparison: Zemaira® vs Placebo; Analysis of the annual rate of change in lung density (TLC+FRC combined) was a linear mixed model with country, inspiration state, time since baseline treatment, and treatment-by-time interaction as fixed effects and participant and participant-by-time interaction as random coefficients at a 1-sided significance level of 0.025; Test type: Superiority or Other; p = 0.029, 95% confidence interval — A 1-sided P-value less than 0.025 and a positive estimate of the treatment difference Zemaira minus placebo (ie, the lower bound of the 95% confidence interval [CI] being greater than zero) will indicate superiority of Zemaira compared with Placebo; Difference in lung density(adjusted P15) = 0.618, 95% CI 2-sided [-0.024 to 1.261] — A mixed model was used to estimate the 95% CI for the difference (Zemaira® - placebo) in annual lung density decline
Statistical Analysis 2: Comparison: Zemaira® vs Placebo; Analysis of the annual rate of change in lung density (TLC) was a linear mixed model with country, time since baseline treatment, and treatment-by-time interaction as fixed effects and participant and participant-by-time interaction as random coefficients at a 1-sided significance level of 0.025; Test type: Superiority or Other; p = 0.017, 95% confidence interval — A 1-sided P-value less than 0.025 and a positive estimate of the treatment difference Zemaira® minus placebo (ie, the lower bound of the 95% CI being greater than zero) will indicate superiority of Zemaira® compared with Placebo; Difference in lung density(adjusted P15) = 0.740, 95% CI 2-sided [0.059 to 1.420] — A mixed model was used to estimate the 95% CI for the difference (Zemaira® - placebo) in annual lung density decline
Statistical Analysis 3: Comparison: Zemaira® vs Placebo; Analysis of the annual rate of change in lung density (FRC) was a linear mixed model with country, time since baseline treatment, and treatment-by-time interaction as fixed effects and participant and participant-by-time interaction as random coefficients at a 1-sided significance level of 0.025; Test type: Superiority or Other; p = 0.090, 95% confidence interval — [p-value comment as in outcome 1, analysis 2]; Difference in lung density(adjusted P15) = 0.478, 95% CI 2-sided [-0.223 to 1.180] — A mixed model was used to estimate the 95% CI for the difference (Zemaira® - placebo) in annual lung density decline

2. Secondary Outcome: Annual Rate of Pulmonary Exacerbations
Description: Primary diagnostic criteria for exacerbations were increased dyspnea, increased sputum volume, and increased sputum purulence. Supporting diagnostic criteria were upper respiratory tract infection, fever without other apparent cause, increased wheezing, and increased cough. For diagnosis, participants had to meet 2 of the 3 primary criteria or 1 primary criterion and 1 supporting criterion. The annual rate was based on the total number of exacerbations and the total number of participant study days for all participants in the specified analysis population and adjusted to 365.25 days.
Time Frame: Over a 2-year period
Population: All participants with A1-PI deficiency who were included in the study and randomized.
Measure: Number (95% Confidence Interval); unit: exacerbations per participant year
Arm/Group | Zemaira® | Placebo
Number analyzed (Participants) | 93 | 87
exacerbations per participant year | 1.70 [1.51 to 1.89] | 1.42 [1.23 to 1.61]

3. Secondary Outcome: Percent Change in FEV1
Description: Percent change from baseline to Month 24.
Time Frame: From baseline to 2 years
Population: All participants with A1-PI deficiency who were included in the study, randomized, and had a baseline and at least one endpoint assessment available.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Zemaira® | Placebo
Number analyzed (Participants) | 89 | 84
percent change | -4.29 (1.26) | -2.06 (1.30)

4. Secondary Outcome: Time to First Pulmonary Exacerbation
Description: Primary diagnostic criteria for exacerbations were increased dyspnea, increased sputum volume, and increased sputum purulence. Supporting diagnostic criteria were upper respiratory tract infection, fever without other apparent cause, increased wheezing, and increased cough. For diagnosis, participants had to meet 2 of the 3 primary criteria or 1 primary criterion and 1 supporting criterion.
Time Frame: Over a 2-year period
Population: All participants with A1-PI deficiency who were included in the study and randomized.
Measure: Median (95% Confidence Interval); unit: Years
Arm/Group | Zemaira® | Placebo
Number analyzed (Participants) | 93 | 87
Years | 0.60 [0.33 to 1.11] | 0.73 [0.46 to 1.17]

5. Secondary Outcome: Change in Lung Density
Description: Change from baseline to Month 24 as measured by centralized, standardized CT lung densitometry. CT scans were acquired at 2 inspiration states: TLC (ie, full inspiration) and FRC (ie, full expiration). Results were adjusted for total lung volume.
Time Frame: From baseline to 2 years
Population: All participants with A1-PI deficiency who were included in the study, randomized, and had a baseline and at least 1 endpoint assessment available.
Measure: Least Squares Mean (Standard Error); unit: g/L
Arm/Group | Zemaira® | Placebo
Number analyzed (Participants) | 80 | 67
g/L
  TLC + FRC combined | -2.33 (0.45) | -3.37 (0.50)
  TLC (N=66 for placebo) | -2.22 (0.47) | -3.54 (0.52)
  FRC | -2.44 (0.50) | -3.33 (0.56)
Statistical Analysis 1: Comparison: Zemaira® vs Placebo; Analysis of the change in lung density (TLC+FRC combined) from baseline to Month 24 was a mixed effects analysis of covariance (ANCOVA) model with country, treatment, and baseline lung density as fixed effects and inspiration state as a repeated random effect at a 1-sided significance level of 0.025; Test type: Superiority or Other; p = 0.058, 95% confidence interval — [p-value comment as in outcome 1, analysis 2]; Difference in lung density(adjusted P15) = 1.04, 95% CI 2-sided [-0.26 to 2.34] — A mixed model ANCOVA was used to estimate the 95% CI for the difference (Zemaira® - placebo) in the change in lung density
Statistical Analysis 2: Comparison: Zemaira® vs Placebo; Analysis of the change in lung density (TLC) from baseline to Month 24 was a mixed effects ANCOVA model with country, treatment, and baseline lung density as fixed effects at a 1-sided significance level of 0.025; Test type: Superiority or Other; p = 0.028, 95% confidence interval — A 1-sided P-value less than 0.025 and a positive estimate of the treatment difference Zemaira® minus placebo (i.e., the lower bound of the 95% CI being greater than zero) will indicate superiority of Zemaira® compared with Placebo; Difference in lung density(adjusted P15) = 1.32, 95% CI 2-sided [-0.03 to 2.67] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Zemaira® vs Placebo; Analysis of the change in lung density (FRC) from baseline to Month 24 was a mixed effects ANCOVA model with country, treatment, and baseline lung density as fixed effects as a repeated random effect at a 1-sided significance level of 0.025; Test type: Superiority or Other; p = 0.115, 95% confidence interval — [p-value comment as in outcome 1, analysis 2]; Difference in lung density(adjusted P15) = 0.89, 95% CI 2-sided [-0.57 to 2.34] — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Change in Exercise Capacity
Description: Exercise capacity was measured as distance walked, using the incremental shuttle walk test. Change from baseline to end of treatment (2 years) in exercise capacity was analysed using an analysis of covariance (ANCOVA).
Time Frame: From baseline to 2 years
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: metre
Arm/Group | Zemaira® | Placebo
Number analyzed (Participants) | 89 | 82
metre | 1.77 (13.0) | 14.86 (13.5)

7. Secondary Outcome: Change in Patient-reported Symptoms
Description: Patient-reported symptoms were measured using the symptoms score component of the St George's Respiratory Questionnaire (SGRQ). SGRQ scores range from 0 to 100, with higher scores indicating more limitations and negative values for change indicating improvement. Change from baseline to end of treatment (2 years) in SGRQ was analysed using an ANCOVA.
Time Frame: From baseline to 2 years
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Zemaira® | Placebo
Number analyzed (Participants) | 85 | 73
units on a scale | -1.19 (1.79) | -0.09 (1.93)

8. Secondary Outcome: Frequency and Intensity of Adverse Events (AEs)
Description: Number of participants with at least one AE, and the number of participants with mild, moderate or severe AEs. AE intensity was defined as mild (does not interfere with routine activities), moderate (interferes with routine activities), or severe (impossible to perform routine activities).
Time Frame: Over a 2-year period
Population: All participants receiving at least 1 infusion of either Zemaira® or placebo.
Measure: Number; unit: participants
Arm/Group | Zemaira® | Placebo
Number analyzed (Participants) | 93 | 87
participants
  At least 1 AE | 92 | 86
  Mild AEs | 13 | 16
  Moderate AEs | 54 | 43
  Severe AEs | 25 | 27

9. Secondary Outcome: Percent Change in Percent Predicted FEV1
Description: Percent change from baseline to Month 24.
Time Frame: From baseline to 2 years
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Zemaira® | Placebo
Number analyzed (Participants) | 89 | 84
percent change | -4.16 (1.27) | -1.90 (1.31)

10. Secondary Outcome: Percent Change in FEV1 Divided by Forced Vital Capacity
Description: Percent change from baseline to Month 24.
Time Frame: From baseline to 2 years
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Zemaira® | Placebo
Number analyzed (Participants) | 89 | 84
percent change | -2.68 (1.36) | 1.56 (1.40)

11. Secondary Outcome: Percent Change in DLCO
Description: Percent change from baseline to Month 24.
Time Frame: From baseline to 2 years
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Zemaira® | Placebo
Number analyzed (Participants) | 89 | 84
percent change | -3.16 (1.96) | -1.85 (2.03)

12. Secondary Outcome: Duration of Pulmonary Exacerbations Relative to Treatment Duration
Description: Defined as the percentage of total treatment duration across participants for 1) exacerbations overall, 2) antibiotic treatment for exacerbations, and 3) hospitalization for exacerbations. Primary diagnostic criteria for exacerbations were increased dyspnea, increased sputum volume, and increased sputum purulence. Supporting diagnostic criteria were upper respiratory tract infection, fever without other apparent cause, increased wheezing, and increased cough. For diagnosis, participants had to meet 2 of the 3 primary criteria or 1 primary criterion and 1 supporting criterion.
Time Frame: Over a 2-year period
Population: All participants with A1-PI deficiency who were included in the study and randomized.
Measure: Mean (Standard Deviation); unit: percentage of total treatment duration
Arm/Group | Zemaira® | Placebo
Number analyzed (Participants) | 93 | 87
percentage of total treatment duration
  Exacerbations (n = 68, 59) | 77.2 (98.8) | 58.9 (109.1)
  Antibiotic treatment (n = 59, 52) | 6.32 (6.75) | 5.55 (6.80)
  Hospitalization (n = 19, 16) | 6.22 (8.79) | 2.16 (1.67)

13. Secondary Outcome: Severity of Pulmonary Exacerbations
Description: Defined as the number of participants requiring 1) antibiotic treatment for exacerbations, and 2) hospitalization for exacerbations. Primary diagnostic criteria for exacerbations were increased dyspnea, increased sputum volume, and increased sputum purulence. Supporting diagnostic criteria were upper respiratory tract infection, fever without other apparent cause, increased wheezing, and increased cough. For diagnosis, participants had to meet 2 of the 3 primary criteria or 1 primary criterion and 1 supporting criterion.
  Antibiotic treatment usage was reported by quarterly interval.
Time Frame: Over a 2-year period
Population: All participants with A1-PI deficiency who were included in the study and randomized.
Measure: Number; unit: participants
Arm/Group | Zemaira® | Placebo
Number analyzed (Participants) | 93 | 87
participants
  Total hospitalizations | 13 | 9
  0 hospitalizations | 80 | 78
  1 hospitalization | 10 | 5
  2 hospitalizations | 1 | 1
  3 hospitalizations | 1 | 3
  >3 hospitalizations | 1 | 0
  Antibiotics: Day 1 to <Month 3 | 22 | 19
  Antibiotics: Month 3 to <Month 6 | 29 | 20
  Antibiotics: Month 6 to <Month 9 | 24 | 15
  Antibiotics: Month 9 to <Month 12 | 21 | 17
  Antibiotics: Month 12 to <Month 15 | 30 | 21
  Antibiotics: Month 15 to <Month 18 | 21 | 15
  Antibiotics: Month 18 to <Month 21 | 26 | 15
  Antibiotics: Month 21 to <Month 24 | 20 | 15

14. Other Pre Specified Outcome: Baseline Lung Density at Total Lung Capacity (TLC) and Forced Residual Capacity (FRC)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Zemaira® | Placebo
Number analyzed (Participants) | 90 | 83
g/L
  TLC | 45.5 (15.8) | 48.9 (15.5)
  FRC | 47.6 (15.7) | 50.7 (15.0)

ADVERSE EVENTS:
Time Frame: For the duration of the study (25 months; 1 month screening period, 24 months treatment period).
Description: The randomized, double-blind investigational product (Zemaira® or placebo) was administered as 60 mg once per week for 24 months. In exceptional cases, a dose of 120 mg could be given to cover a 2-week period. The safety population comprised all participants receiving at least 1 infusion of either Zemaira® or placebo.
Arm/Group | Zemaira® | Placebo
Serious Adverse Events (participants affected / at risk) | 28/93 | 28/87
Other Adverse Events (participants affected / at risk) | 90/93 | 84/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zemaira® (N=93) | Placebo (N=87)
Pneumonia (Infections and infestations) | 3 (3) | 4 (6)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 4 (5)
Diverticulitis (Infections and infestations) | 1 (1) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Graft infection (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 9 (18) | 2 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Adhesion (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Condition aggravated (General disorders) | 1 (2) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Aortic aneurysm repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Tonsillectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Transurethral prostatectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Eye inflammation (Eye disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zemaira® (N=93) | Placebo (N=87)
Nasopharyngitis (Infections and infestations) | 30 (54) | 26 (61)
Lower respiratory tract infection (Infections and infestations) | 18 (88) | 17 (68)
Upper respiratory tract infection (Infections and infestations) | 15 (28) | 14 (26)
Influenza (Infections and infestations) | 14 (14) | 10 (12)
Sinusitis (Infections and infestations) | 12 (17) | 11 (19)
Bronchitis (Infections and infestations) | 12 (25) | 10 (15)
Pneumonia (Infections and infestations) | 8 (12) | 10 (19)
Urinary tract infection (Infections and infestations) | 8 (12) | 6 (9)
Gastroenteritis (Infections and infestations) | 4 (5) | 6 (6)
Rhinitis (Infections and infestations) | 7 (8) | 3 (3)
Pharyngitis (Infections and infestations) | 4 (5) | 5 (8)
Respiratory tract infection (Infections and infestations) | 1 (2) | 8 (12)
Tooth abscess (Infections and infestations) | 1 (1) | 5 (5)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 27 (93) | 19 (53)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 22 (36) | 10 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (33) | 8 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 (28) | 8 (9)
Condition aggravated (General disorders) | 20 (62) | 14 (41)
Fatigue (General disorders) | 8 (14) | 10 (12)
Pyrexia (General disorders) | 12 (14) | 6 (8)
Oedema peripheral (General disorders) | 6 (6) | 10 (14)
Influenza like illness (General disorders) | 4 (5) | 5 (5)
Chest pain (General disorders) | 5 (5) | 1 (1)
Headache (Nervous system disorders) | 38 (101) | 34 (108)
Dizziness (Nervous system disorders) | 6 (13) | 8 (8)
Nausea (Gastrointestinal disorders) | 14 (22) | 8 (11)
Abdominal pain upper (Gastrointestinal disorders) | 9 (11) | 6 (11)
Diarrhoea (Gastrointestinal disorders) | 8 (9) | 7 (9)
Toothache (Gastrointestinal disorders) | 5 (7) | 9 (10)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (5) | 5 (5)
Vomiting (Gastrointestinal disorders) | 5 (10) | 5 (6)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 6 (8)
Gastritis (Gastrointestinal disorders) | 6 (9) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 9 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (9) | 6 (9)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 (10) | 4 (7)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6) | 4 (5)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 5 (5)
Hypertension (Vascular disorders) | 6 (6) | 10 (10)
Anxiety (Psychiatric disorders) | 5 (12) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements and restrictions on publishing may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.